CLINICAL TRIAL: NCT03958370
Title: Validation of Consumer Activity Monitors in Postoperative Total Arthroplasty Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Benaroya Research Institute (Other)
Collaborators: Virginia Mason Hospital/Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: IRB17-053
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Arthropathy of Knee; Arthritis Knee; Arthritis, Degenerative
Keywords: Fitbit; Activity Monitor; Step Count; Total Knee Replacement; Arthroplasty
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fitbit
  Interventions: Other: Fitbit

INTERVENTIONS:
Other: Fitbit — Fitbit use during physical therapy session

SUMMARY:
Mobilization and rehabilitation are essential components of a successful functional recovery following total hip and knee arthroplasties. Currently, we have no good measure of how mobile patients are after their surgery. Recent technological advances in personal activity monitors, such as the Fitbit, might provide medical providers and patients the opportunity to more objectively monitor their postoperative mobility and recovery course. However, these consumer activity monitors have yet to be validated in terms of their accuracy and utility for monitoring mobility in the immediate postoperative setting in arthroplasty patients. Our goal is to validate one of the most popular consumer activity monitors, the Fitbit Zip, in the postoperative total joint arthroplasty patient population.

DETAILED DESCRIPTION:
Early mobilization following total hip and knee arthroplasty surgeries is important in decreasing the risk of complications such as deep venous thrombosis, pulmonary embolus, pneumonia, and urinary retention. It is also generally accepted that early mobilization may help prevent late complications such as joint stiffness or arthrofibrosis. Aside from these complications, patient satisfaction and length of hospital stay both seem to be correlated with early mobilization with poor mobility negatively impacting both outcomes. Therefore, it is important for clinicians to ensure that patients are adequately mobilizing in the immediate postoperative period to promote a successful recovery after total hip or knee arthroplasty.

Consumer activity monitors are generally manufactured to be used in a relatively healthy, ambulatory population. Their accuracy has been validated in multiple studies in healthy subjects in a variety controlled settings. Based on these validity studies, it is clear that some of these consumer activity monitors have worse accuracy in certain situations, such as slower-paced walking or in people using assistive devices for ambulation, such as canes. The limitations of these devices in these settings could be problematic for monitoring post-arthroplasty patients since all these patients ambulate slowly, with an altered gait, and with a walker. No studies to date have looked at the accuracy of consumer activity monitors in the immediate postoperative arthroplasty population.

The consumer activity monitor market is rapidly evolving and changing, so much so that monitors used just last year might be obsolete this year. Therefore, rather than examining the accuracy of one device versus another, it is more applicable to determine what location is most accurate for placement of these monitors to help providers counsel patients on proper use postoperatively.

Our goal for this study is to validate and to determine the best location for placement of the Fitbit Zip in the postoperative total joint arthroplasty patient population.

ELIGIBILITY:
Inclusion Criteria:

* primary unilateral total knee arthroplasty
* ASA class I-IV
* expected to ambulate with PT on postoperative day 1 or 2
* no history of chronic opioid or alcohol use
* no history of delirium
* ability to read and understand English
* patient agreement

Exclusion Criteria:

* patient refusal,
* bilateral arthroplasty patients,
* patients who are non- ambulatory preoperatively (e.g. wheelchair bound),
* patients who are not expected to ambulate with PT either due to intraoperative or postoperative complications,
* patients with contact precautions

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any person who is over 18 years old, a procedural candidate (having a total arthroplasty surgery at Virginia Mason Medical Center), and can understand English sufficiently to consent for the study can be included
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Step Count Obtained from Fitbit | Postoperative day 0-2
  Comparing Fitbit step counts to observer counted steps during physical therapy sessions during inpatient stay

SECONDARY OUTCOMES:
Correlation of Step Count to Distance and Time Ambulated | Postoperative day 0-2
  See if Fitbit counts are more or less accurate depending on distance and time ambulated

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No